CLINICAL TRIAL: NCT00196547
Title: Randomized Placebo-controlled Trial of Montelukast in Modulating Exacerbations of Asthma in Children, September 2005
Brief Title: Montelukast in Modulating Exacerbations of Asthma in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Firestone Institute for Respiratory Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R.P. #05-2440
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: Asthma; Respiratory viral infections; Exacerbations; Pediatric; Leukotriene receptor antagonists; School
MeSH Terms: conditions — Asthma | interventions — montelukast; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Montelukast (drug)

SUMMARY:
The purpose of the study is to determine if Montelukast added to other therapy, if any, will reduce the severity of asthma symptoms in children during the high incidence of respiratory viral infections that occur in children in the post Labor Day school return period.

DETAILED DESCRIPTION:
Between 1990- and 2003, we identified in Ontario, and subsequently across Canada, a striking increase in hospital admissions for asthma in children occurring predictably in the third week of September every year.1 In 2000 we undertook a retrospective case-control study comparing the clinical characteristics of children using local emergency rooms for asthma in September, with those of children presenting during the non-epidemic months of July-August. Based on that pilot study of 169 children, we developed a larger prospective case-control study of clinical and biological characteristics of children recruited as they presented to an emergency room for asthma during September 2001. The control group for this study were children recruited from the community who had symptomatic asthma but did not have a September exacerbation requiring emergency room utilization. We identified the presence of rhinovirus in the majority of children attending an ER with acute asthma, and also found rhinovirus in a substantial proportion of the community based controls. We also found a highly significant difference in use of medications for asthma, with the ER cases being much less likely to be receiving adequate anti-inflammatory medication. In September 2004 we conducted a pilot randomized controlled blinded clinical trial of the efficacy of montelukast in reducing morbidity caused by asthma exacerbations associated with respiratory viral infections (RVI) in children aged 2 to 14. We found a highly significant reduction in reported symptom free days in the montelukast group. The current study is a randomized placebo-controlled trial of montelukast, during September 2005 to confirm the results of our pilot study and to examine the effectiveness of montelukast in reducing asthma morbidity during RVIs in different age and sex groups with a range of risk of exacerbations. We also wish to compare the effectiveness of montelukast to placebo in reducing asthma morbidity during RVIs between groups of children concurrently taking no or other classes of asthma control medications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-14 years inclusive
* Doctor-diagnosed asthma
* Needing a beta-agonist inhaler at least once weekly on average for symptom relief
* At least one day lost from school in the past year, or significantly limited activity, because of asthma
* A history of asthma exacerbations associated with apparent respiratory viral infections
* Parent or guardian who is willing to provide informed consent
* Willing to give assent

Exclusion Criteria:

* Non-English speaking
* Unable to understand purpose of study and give consent
* Concomitant respiratory or other major illness e.g. cystic fibrosis, cardiac disease
* Currently using montelukast or other leukotriene receptor antagonist
* Using regular oral corticosteroid
* An asthma exacerbation requiring medical intervention during August 2005

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2005-09; Study Completion 2005-11

PRIMARY OUTCOMES:
Daily asthma symptom score

SECONDARY OUTCOMES:
Unscheduled physician visits (including ER)
Oral-cortico-steroid use

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm R Sears, MB. ChB, Principal Investigator — Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton; Neil W Johnston, MSc, Study Director — Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton
Locations (1):
- Firestone Institute for Respiratory Health, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Johnston NW, Johnston SL, Duncan JM, Greene JM, Kebadze T, Keith PK, Roy M, Waserman S, Sears MR. The September epidemic of asthma exacerbations in children: a search for etiology. J Allergy Clin Immunol. 2005 Jan;115(1):132-8. doi: 10.1016/j.jaci.2004.09.025. PMID 15637559
- [Background] Bisgaard H, Zielen S, Garcia-Garcia ML, Johnston SL, Gilles L, Menten J, Tozzi CA, Polos P. Montelukast reduces asthma exacerbations in 2- to 5-year-old children with intermittent asthma. Am J Respir Crit Care Med. 2005 Feb 15;171(4):315-22. doi: 10.1164/rccm.200407-894OC. Epub 2004 Nov 12. PMID 15542792
- [Derived] Johnston NW, Mandhane PJ, Dai J, Duncan JM, Greene JM, Lambert K, Sears MR. Attenuation of the September epidemic of asthma exacerbations in children: a randomized, controlled trial of montelukast added to usual therapy. Pediatrics. 2007 Sep;120(3):e702-12. doi: 10.1542/peds.2006-3317. PMID 17766511